CLINICAL TRIAL: NCT03170453
Title: Cognitive Enhancement Therapy for Adult Autism Spectrum Disorder
Brief Title: Confirmatory Efficacy Trial of Cognitive Enhancement Therapy for Adult Autism Spectrum Disorder
Acronym: PerspectivesII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Shaun M. Eack, Professor of Social Work and Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19080150; R01MH106450 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-05-31 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-06

CONDITIONS: Autistic Disorder; Autism Spectrum Disorder; Asperger Syndrome; Pervasive Developmental Disorder
Keywords: Autism; Autism Spectrum Disorder; Asperger's Syndrome; Pervasive Developmental Disorder; Cognition; Social Cognition; Psychosocial Treatment; Cognitive Enhancement Therapy; Enriched Supportive Therapy; Therapy; Psychotherapy
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Asperger Syndrome; Child Development Disorders, Pervasive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Enhancement Therapy (Experimental): This research treatment aims to help with problems in thinking, planning, and socialization. Participants begin with cognitive training using computer software programs. They also participate in a small social-cognitive group to learn about their condition and how to act wisely in social situations by developing the abilities needed to understand another person's perspective, evaluate social contexts, and be foresightful.
  Time commitment: about 3½ hours per week; Location: Pittsburgh, PA only
  Interventions: Behavioral: Cognitive Enhancement Therapy
- Enriched Supportive Therapy (Active Comparator): This research treatment uses individual supportive therapy to help adults learn about autism spectrum disorder, manage their emotions and stress, improve their social skills, and cope with everyday problems. Participants will learn about the impact of stress on their lives, and how to identify their own early cues of distress and apply effective coping strategies.
  Time commitment: about 1 hour per week; Location: Pittsburgh, PA only
  Interventions: Behavioral: Enriched Supportive Therapy

INTERVENTIONS:
Behavioral: Cognitive Enhancement Therapy — An 18-month comprehensive, small group approach for the remediation of cognitive deficits in neurodevelopmental disorders consisting of individual sessions and 45 group training sessions in social cognition that are integrated with approximately 60 hours of computer assisted training in attention, memory, and problem solving skills.
  Arms: Cognitive Enhancement Therapy
Behavioral: Enriched Supportive Therapy — An 18-month intervention that uses individual supportive therapy to help adults learn about autism spectrum disorder, manage their emotions and stress, improve their social skills, and cope with everyday problems. Participants will learn about the impact of stress on their lives, and how to identify their own early cues of distress and apply effective coping strategies.
  Arms: Enriched Supportive Therapy

SUMMARY:
This study will investigate and confirm the efficacy of two psychological treatments for adults with autism spectrum disorder. Cognitive Enhancement Therapy (CET) is a cognitive remediation intervention that aims to help adults with problems in thinking, planning, and socialization. Enriched Supportive Therapy (EST) is an individual supportive therapy that aims to help adults learn about their condition, manage their emotions and stress, improve their social skills, and cope with everyday problems.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is characterized by marked impairments in social and non-social cognitive ability that persist well into adulthood and contribute to significant functional disability. The treatment of ASD has focused almost exclusively on children, and few empirically supported interventions are available to address the core cognitive and functional challenges individuals with ASD face as they transition to adulthood. This study will investigate and confirm the efficacy of two psychological treatments for adults with autism spectrum disorder. Cognitive Enhancement Therapy (CET) is a cognitive remediation intervention that aims to help adults with problems in thinking, planning, and socialization. Enriched Supportive Therapy (EST) is an individual supportive therapy that aims to help adults learn about their condition, manage their emotions and stress, improve their social skills, and cope with everyday problems.

Participation in this study will last 30 months. Potential participants must be able to attend weekly treatment sessions in Pittsburgh, PA.

The study design is a 30-month (2.5 years) randomized-controlled confirmatory efficacy trial, where eligible participants will be randomized to the CET or EST study treatments. Participants will be treated with the study interventions for 18 months, and then followed for 12 additional months to assess the lasting impact of the study interventions. All participants will complete cognitive, clinical, and neuroimaging (magnetic resonance imaging) assessments prior to starting the study treatments and then at specified intervals thereafter to evaluate the impact of the study treatments on cognition, adaptive function, and the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-45 years
* Diagnosis of autism, Asperger's syndrome, or pervasive developmental disorder not otherwise specified (NOS) verified by the autism diagnostic observation schedule (ADOS) or autism diagnostic interview-revised (ADI-R)
* Presence of significant social and cognitive disability, based on the Cognitive Style and Social Cognition Eligibility Interview (Hogarty et al., 2004)
* Intelligence quotient (IQ) greater than 80
* Ability to read and speak fluent English
* Availability of a family member or close friend allowed to provide information on the participant
* Ability to attend weekly treatment sessions in Pittsburgh, PA

Exclusion Criteria:

* Organic brain syndrome
* IQ < 80
* English language skills below a sixth grade level
* Persistent suicidal or homicidal behavior
* History of substance abuse or dependence within the past 3 months
* Comorbid attention deficit hyperactivity disorder (ADHD) that is untreated
* Comorbid personality disorder
* History of disruptive or violent behavior
* Any magnetic resonance imaging contraindications

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Neurocognition | Pre-treatment, 9, 18, and 30 months
  Composite measure of neuropsychological tests designed to assess neurocognitive function. Multiple measures will be aggregated into a composite index by scaling measures to common (z) metric, reverse coding relevant items, and computing their average to provide a single composite score for this outcome.
Change in Social cognition | Baseline, 9, 18, and 30 months
  Composite measure of performance-based and interview tests designed to assess social-cognitive function. Multiple measures will be aggregated into a composite index by scaling measures to common (z) metric, reverse coding relevant items, and computing their average to provide a single composite score for this outcome.

SECONDARY OUTCOMES:
Change in Functional outcome | Baseline, 9, 18, and 30 months
  Composite measure of interview assessments of social, vocational, interpersonal, independent living, and other domains of functional outcome. Multiple measures will be aggregated into a composite index by scaling measures to common (z) metric, reverse coding relevant items, and computing their average to provide a single composite score for this outcome.

OTHER OUTCOMES:
Change in Processing Speed/Attention | Baseline and 3 months
  Standardized neuropsychological tests of processing speed and attention. Multiple measures will be aggregated into a composite index by scaling measures to common (z) metric, reverse coding relevant items, and computing their average to provide a single composite score for this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun M Eack, Ph.D., Principal Investigator — University of Pittsburgh; Nancy J Minshew, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the National Database for Autism Research
Time Frame: Final data will be deposited to NDAR upon study completion.
Access Criteria: Access will be available to qualified investigators and institutions who are eligible for access to NDAR.